CLINICAL TRIAL: NCT01732055
Title: Partner-Assisted Interpersonal Psychotherapy or Antidepressant Medication for Antenatal Depression
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study ended because recruitment goals unmet and further funding unlikely
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Foundation of Hope for Research and Treatment of Mental Illness (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0235
Record Dates: First submitted 2012-11-06; First posted 2012-11-22 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Partner Assisted Interpersonal Psychotherapy; Treatment as Usual
Keywords: Pregnancy; Antenatal; Major Depressive Disorder; Psychotherapy; Antidepressant Medication; Partners; Spouses; Interpersonal Psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics; Watchful Waiting; Antidepressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partner-Assisted Interpersonal Psychotherapy (Active Comparator): Partner-Assisted Interpersonal Psychotherapy is an 8-week series of psychotherapy sessions attended by the patient and her identified partner.
  Interventions: Behavioral: Partner-Assisted Interpersonal Psychotherapy
- Treatment as Usual (Other): Treatment prescribed for subjects by the UNC Perinatal Psychiatry clinic physicians according to the clinic algorithm.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Partner-Assisted Interpersonal Psychotherapy
  Other Names: PA-IPT; PAT
  Arms: Partner-Assisted Interpersonal Psychotherapy
Other: Treatment as Usual — Because treatment(s) are prescribed for subjects by the UNC Perinatal Psychiatry physicians, it is impossible for the investigators to list each potential medication and dosage that might be prescribed to women randomized to this condition. The medication regimens are individual, and some women may opt against medication altogether (and still be eligible to enroll). Women who refuse antidepressant medication will attend visits at the same intervals as those in the study arms for evaluation of safety and symptoms.
  Other Names: TAU; Watchful Waiting; Antidepressant Medication
  Arms: Treatment as Usual

SUMMARY:
Purpose: To compare a novel psychotherapy, Partner-Assisted Interpersonal Psychotherapy (PA-IPT), with treatment as usual (TAU) in a sample of pregnant women seeking treatment for Major Depressive Disorder (MDD) at the University of North Carolina at Chapel Hill (UNC-CH) Perinatal Psychiatry Program.

Participants: 52 women, ages 18-45, who are 16-29 weeks pregnant and experiencing a depressive episode, and their partners.

Methods: Women and their identified partners will complete a diagnostic interview, complete measures of depressive symptom severity at baseline, and be randomized to treatment with PA-IPT or TAU. Women randomized to TAU will be treated by UNC physicians according to the UNC-CH Perinatal Psychiatry Program's algorithm for treatment of prenatal MDD (usually one of a number of antidepressant medications, tailored to the individual, although some women may opt against medication altogether and still be eligible to enroll). Women randomized to PA-IPT will participate in 8 therapy sessions with their identified partner over a 12-week period, along with one refresher session at or around 6 weeks postpartum. Women and partners will be assessed for change in depressive symptoms and relationship satisfaction during pregnancy at visits 4 and 8, and postpartum at 6-week and 6-month visits.

Hypothesis: The investigators anticipate notable improvement in both groups similar in magnitude, however it is hypothesized that couples participating in PA-IPT will have higher relationship satisfaction post-treatment (controlling for baseline satisfaction) than those receiving TAU.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-45 years
* 16-29 weeks estimated gestational age
* Able to provide informed consent
* English or Spanish language literacy
* In a committed relationship cohabiting for at least 6 months with a Dyadic Adjustment Scale rating < 90 or with an identified family member or friend residing in the same home
* Meet criteria for Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition Text Revision (DSM-IV) diagnosis of Major Depressive Disorder (MDD)
* HRSD-17 score is equal or greater than 16 at diagnostic evaluation and randomization
* Medically healthy and without fetal anomaly according to history

Exclusion Criteria:

* No identified primary care, nurse midwife, or obstetrical physician to monitor pregnancy; participant or physician refuses to sign release of information
* By patient report, history of partner verbal, emotional, or physical abuse
* Partner unable or unwilling to participate
* DSM-IV diagnoses of bipolar 1 or 2 or any psychotic episode
* Substance abuse within the last 6 months
* Eating Disorder
* Current use of other therapies for depression including individual psychotherapy, herbal remedies or other complementary/alternative therapies, antidepressant medication outside the study protocol
* Active suicidal ideation
* Identified partner has DSM-IV diagnoses of bipolar 1 or 2 or any psychotic episode
* Interpersonal violence or abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression-17 item version (HRSD-17) | Baseline (16-29 weeks pregnancy) until Endpoint (6 months postpartum)
  Change from baseline in symptoms of Major Depressive Disorder

SECONDARY OUTCOMES:
Dyadic Adjustment Scale (DAS) | Baseline (16-29 weeks pregnancy) until Endpoint (6 months postpartum)
  Change from baseline in relationship satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Anna R. Brandon, PhD, MSCS, Principal Investigator — University of North Carolina, Chapel Hill; Samantha Meltzer-Brody, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals and Clinics, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Brandon AR, Ceccotti N, Hynan LS, Shivakumar G, Johnson N, Jarrett RB. Proof of concept: Partner-Assisted Interpersonal Psychotherapy for perinatal depression. Arch Womens Ment Health. 2012 Dec;15(6):469-80. doi: 10.1007/s00737-012-0311-1. Epub 2012 Oct 4. PMID 23053218